CLINICAL TRIAL: NCT02748161
Title: Surefire vs. Endhole for DEB-TACE: Quantifying Hepatic Artery Embolization to Improve Outcomes by Comparing Two Different Catheter Systems for DEB-TACE (QED Study)
Brief Title: DEB-TACE for Hepatocellular Carcinoma
Acronym: QED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Surefire Medical, Inc. (Industry)
Responsible Party: Sponsor
Organization: SurefireMedical (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00061366
Record Dates: First submitted 2016-04-18; First posted 2016-04-22 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; DEB-TACE; QED
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DEB-TACE: Standard Endhole Catheter (Active Comparator): Subjects will undergo DEB-TACE using a standard endhole catheter.
  Interventions: Procedure: DEB-TACE
- DEB-TACE: Surefire Infusion System (Active Comparator): Subjects will undergo DEB-TACE using the Surefire Infusion System.
  Interventions: Procedure: DEB-TACE

INTERVENTIONS:
Procedure: DEB-TACE — Transarterial chemoembolization with doxorubicin-eluting beads.

SUMMARY:
Patients enrolled in this study have been diagnosed with hepatocellular carcinoma (HCC) and are scheduled to have a procedure called drug-eluting bead trans-arterial chemoembolization (DEB-TACE). During the DEB-TACE procedure, very small beads are mixed in with a chemotherapy drug, doxorubicin, and delivered to the tumor through an arterial catheter.

The DEB-TACE procedure allows the treatment to be delivered directly into the liver. It also causes arterial embolization, the process in which a blood vessel is blocked. Treatment of HCC using DEB-TACE may help delay tumor progression and can downstage (decrease the size) the cancer in order to meet the criteria which may allow patients to become candidates for liver transplantation. The purpose of this study is to compare tumor response and medical outcomes for patients who undergo DEB-TACE with standard endhole catheter versus Surefire® Infusion System.

DETAILED DESCRIPTION:
Conventional transarterial chemoembolization with lipiodol/doxorubicin (cTACE) is known to prolong survival compared to supportive therapy in certain patients with unresectable HCC, including patients with unilateral portal vein invasion (PVI). TACE with doxorubicin-eluting beads (DEB-TACE) is a relatively new modality associated with favorable systemic doxorubicin exposure/toxicity and liver-specific toxicity compared to cTACE and studies have documented its safety and efficacy. DEB-TACE is currently utilized for: (1) patients who have unresectable HCC; and (2) patients who meet the Milan Criteria and currently on liver transplantation lists.

The biggest challenge for these procedures has been the inability to actually quantify embolization in a real-time setting to provide immediate feedback to the operator. Although various methods, such as perfusion analysis with CT or MRI, have been described, these require advanced imaging equipment/capabilities, extensive post processing analysis, and can create challenging workflows.

Currently the best results occur when the dose is delivered in a highly targeted manner into the tumor. Dense accumulation of embolic spheres or lipiodol into the tumor as documented by CT has been shown to have improved outcomes. However, with standard endhole catheters achieving maximum delivery of embolic agents is limited by the development of stasis and subsequent non-target injury.

As DEB-TACE is performed through an endhole catheter with either stasis or substasis as an endpoint. The current methodology is extremely subjective, lacks a quantifiable endpoint, and results in various degrees of embolization on patients. Often this can result in repeat procedures or the progression of tumor.

Recently, there has been FDA clearance of a new anti-reflux catheter, Surefire® Infusion System (SIS, Westminster, CO). The current design has an expandable tip which collapses during forward flow, and then dynamically seal off the vessel with reversal of flow, analogous to a valve. SIS, with its expandable tip microcatheter, has been demonstrated clinically to cause a slight decrease in intra-arterial pressure in the antegrade, or downstream, vascular compartment. Although this device was designed primarily to prevent retrograde reflux of embolic agents, the downstream blood pressure reduction may serve as a biomarker on quantifying embolization.

The goal is to develop a method that: (1) allows maximum delivery of embolic spheres into the tumor tissue to stasis without reflux; (2) enables direct real time numerical quantification on the degree of embolization; and (3) provides an intra-procedural functional parameter which could be used to guide the optimal therapeutic endpoints at the time of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, inclusive
* Diagnosis of HCC
* Meets UCSF criteria: a single lesion less than or equal to 6.5 cm in diameter or 2-3 lesions less than or equal to 4.5 cm with total tumor diameter less than or equal to 8 cm.
* No portal invasion or extrahepatic spread on imaging.
* Child-Pugh Class A or B.
* No previous chemotherapy, radiotherapy or transarterial embolization (with or without chemotherapy).
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* A discrete hepatic artery feeding the tumor with diameter of the vessels equal to or greater than 1.5 mm.

Exclusion Criteria:

* Bilirubin levels greater than 3 mg/dl
* AST or ALT greater than 5 times upper limit of normal or greater than 250 U/l.
* Advanced tumoral disease (vascular invasion or extrahepatic spread, portal vein thrombosis of bland or malignant origin), or diffuse HCC, defined as 50% liver involvement).
* Contraindications for doxorubicin administration.
* Subject has a known history contraindicating contrast dye or iodine that cannot be safely controlled via antihistamine, steroids, or with any other agent.
* Unable or unwilling to provide informed consent.
* Vessels providing flow to the tumor that are less than 1.5 mm in diameter.
* Women who are pregnant or breast feeding.
* Women of childbearing potential who are not using an acceptable method of birth control (e.g., pill, patch, IUD, ring, condom, sponge, foam).
* Portal vein thrombosis of bland or malignant origin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Objective tumor response | 1 month following initial DEB-TACE procedure

SECONDARY OUTCOMES:
Objective tumor response | 3 months following initial DEB-TACE procedure (or 1 month following retreatment if DEB-TACE retreatment performed)
Dose of doxorubicin-eluting beads used during DEB-TACE procedure(s) | Procedure
Number of repeat DEB-TACE procedures per lesion | 3 months following initial DEB-TACE procedure

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Phoenix, Arizona
  - UCLA, Los Angeles, California
  - USC, Los Angeles, California
  - Radiology Imaging Associates, Denver, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - University of Maryland, Baltimore, Maryland
  - New York University, New York, New York
  - Cleveland Clinical Foundation, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No